CLINICAL TRIAL: NCT04828447
Title: Recipe for Heart Health: A Plant-Based Culinary Diet Intervention to Test Independent Benefits of Olive Oil
Brief Title: Recipe for Heart Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Recipe for Heart Health; IRB202002194 (Other: UF IRB-01)
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: Pilot prospective randomized crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Olive Oil (Experimental): There will be a total of 4 in-person clinic visits as well as 8 weekly remote cooking classes and individual sessions with a registered dietitian. Subject will first have a physical exam, have their blood (about 3 tablespoons) and urine collected, complete surveys, and talk about their eating style and meal planning. Subject will then follow a plant-based diet high in olive oil for 4 weeks before switching to the other type of diet for 4 weeks.
  Interventions: Dietary Supplement: Olive Oil
- Low Olive Oil (Experimental): There will be a total of 4 in-person clinic visits as well as 8 weekly remote cooking classes and individual sessions with a registered dietitian. Subject will first have a physical exam, have their blood (about 3 tablespoons) and urine collected, complete surveys, and talk about their eating style and meal planning. Subject will then follow a plant-based diet low in olive oil for 4 weeks before switching to the other type of diet for 4 weeks.
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Olive Oil — Subjects will be randomized to either high or low dose of olive oil and follow a whole food plant based diet.

SUMMARY:
The overall objectives of this project are to compare clinical parameters in moderate risk Atherosclerotic Cardiovascular Disease (ASCVD) patients following a Whole Food Plant Based (WFPB) diet containing a high (4 TB) compared to a low (<1 tsp) amount of raw extra virgin olive oil.

DETAILED DESCRIPTION:
Up to sixty-eight primary prevention outpatient adults with intermediate to high ASCVD risk factors will be randomized in a crossover fashion to follow a WFPB diet without animal products that is either high (4 tablespoons) or low (< ~1 teaspoon) in raw extra virgin olive oil. After confirming eligibility and patients provide consent, the research team will randomize the participant at the baseline visit. The baseline visit and run-in visit 1 will follow as described below. With the intent of recruiting cohorts of ten, a group of participants will subsequently begin the first Whole Food Plant Based culinary diet intervention for four weeks, followed by a one-week (+ 3 days) washout period before switching to the opposite oil diet for an additional four weeks. During each of the 4-week interventions, participants will attend weekly cooking sessions that align with the dietary intervention with a registered dietitian. Patients will be asked to maintain levels of physical activity through the duration of the study. Data will be collected at the patient's cardiology visits before and after each diet intervention for a total of four in-person visits excluding the screening visit.

ELIGIBILITY:
Inclusion Criteria:

-Adult patients with borderline to high risk for ASCVD

Exclusion Criteria:

-Adult patients with known cardiovascular disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Low Density Lipoprotein-Cholesterol | 4 weeks
  Change from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Monica Aggarwal, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krenek AM, Mathews A, Guo J, Courville AB, Pepine CJ, Chung ST, Aggarwal M. Recipe for Heart Health: A Randomized Crossover Trial on Cardiometabolic Effects of Extra Virgin Olive Oil Within a Whole-Food Plant-Based Vegan Diet. J Am Heart Assoc. 2024 Aug 6;13(15):e035034. doi: 10.1161/JAHA.124.035034. Epub 2024 Jul 24. PMID 39045758